CLINICAL TRIAL: NCT01049568
Title: A Pilot Study Using Cell Phone Interactions to Improve Medication Adherence in Adolescents Who Have Previously Failed Antiretroviral Therapy Due to Non-Adherence
Brief Title: Cell Phone Reminders Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATN 078
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-03

CONDITIONS: HAART Non-Adherence; HIV; HIV Infections
Keywords: HIV; Cell phone; HAART
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cell Phone Intervention (Experimental)
  Interventions: Behavioral: Cell Phone Intervention
- Control (No Intervention): Control group participants will participate in all on-study evaluations, except the intervention exit interviews.
  Data will be collected using the ACASI and CRFs at entry, weeks 6, 12, 24, 36, 48 and the premature discontinuation visits. Measures will assess social support, coping, self-efficacy, substance use, adherence, life stressors, perceived stress, psychological symptoms and health service utilization.

INTERVENTIONS:
Behavioral: Cell Phone Intervention — Cell phone support, including reminders, assessment of barriers to adherence, problem solving and referrals conducted by an Adherence Facilitator.
  Data will be collected using the ACASI and CRFs at entry, weeks 6, 12, 24, 36, 48 and the premature discontinuation visits. Measures will assess social support, coping, self-efficacy, substance use, adherence, life stressors, perceived stress, psychological symptoms and health service utilization.
  Arms: Cell Phone Intervention

SUMMARY:
This study will use a longitudinal, experimental design. Participants will be randomized to either the intervention or the control group.

The intervention will involve cell phone support, including reminders, assessment of barriers to adherence, problem solving and referrals conducted by an Adherence Facilitator.

Control group participants will participate in all on-study evaluations, except the intervention exit interviews.

DETAILED DESCRIPTION:
Forty participants, non-adherent to HAART at study start, will be randomly assigned to either a 1) "Cell Phone Adherence Facilitator" group (intervention group) or a 2) control group. In the intervention group, a Cell Phone Adherence Facilitator will initiate a short (typically five minutes or less) contact Monday through Friday (excluding major holidays) with each participant to enhance their adherence to HAART. Occasionally, calls may be longer if crises arise that can be addressed by the Adherence Facilitator. Calls from the Adherence Facilitator will occur once or twice a day (depending on dosing schedule) and go on for 24 weeks in the intervention group. Calls will occur at a time soon after the prescribed dose is supposed to be taken, but also one convenient to the participant and the Adherence Facilitator.

All participants regardless of condition will be followed for 48 weeks. This intervention will be examined as a tool to address participant-specific, healthcare systems and participant-provider relationship barriers to ARV adherence.

ELIGIBILITY:
Inclusion Criteria:

Documented HIV-positive infected either behaviorally or perinatally as determined by medical record review or verbal verification from referring professional.

Age 15 and 0 days to 24 years and 364 days. Enrolled in care at an AMTU or affiliated site.

History of non-adherence to one or more components of antiretroviral therapy, defined as meeting one of the following criteria:

* Currently prescribed HAART and reports to care provider less than 90% adherence in previous month and has viral load greater than 1000 copies/ml when last evaluated (within the last four weeks);
* Discontinued HAART in the past while documented to be less than 90% adherent during the most recent antiretroviral treatment; and
* Agreed to initiate antiretroviral treatment in the past, but never initiated. Able to speak and understand English. Willing to provide informed consent or assent.

Exclusion Criteria:

Evidence of cognitive impairment or other mental condition (including substance abuse) that limits his/her ability to complete intervention and assessments (per PI or designee discretion). Participants with stable and treated mental health/substance abuse disorders are acceptable for inclusion with protocol team approval.

Any condition, including active substance abuse that is expected to limit the likelihood that the participant may maintain involvement for the entire year on-study (per PI or designee discretion with protocol team approval).

No participant consent, parental permission or youth assent (as appropriate). Minors unable to acquire parental/guardian consent, even if not living at home, will not be able to participate as a change in housing status during the study might require premature discontinuation.

Current participation in another behavioral interventional trial.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To examine the content of the Adherence Facilitator's conversation; including reported stressful life circumstances, what solutions were offered, and acceptability of the intervention among intervention participants. | 1 year
To examine the trends of therapeutic success at 6 and 12 months, as measured by lowered viral load, and self-reported adherence among intervention versus control group participants. | 1 year

SECONDARY OUTCOMES:
To examine the trends of self-reported and chart-documented service utilization among intervention versus control participants. | 1 year
To identify the characteristics of youth who may require longer-term adherence support with cell phone conversations based on their self-reported scores of depression, life stressors, substance use, and their utilization of services. | 1 year
To track the costs of implementation of cell phone contacts with Adherence Facilitators in the adolescent clinical setting by collecting the monthly cost of youths' cell phones. | 1 year
To evaluate barriers to and promoters of implementation of cell phone support through qualitative interviews with intervention participants and Adherence Facilitators. | 1 year
To examine the trends for self-reported adherence self-efficacy, perceived stress, and problem-solving orientation towards medication among intervention versus control group participants. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Belzer, MD, Study Chair — Adolescent Trials Network
Locations (5):
- United States (5):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - Tulane University Health Sciences Center, New Orleans, Louisiana

REFERENCES:
- See also: ATN Website — http://www.atnonline.org